CLINICAL TRIAL: NCT04793737
Title: Precision Radiation of Immune Checkpoint Therapy Resistant Melanoma Metastases
Acronym: PROMMEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Hildur Helgadottir, Principal Investigator, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROMMEL
Record Dates: First submitted 2021-02-17; First posted 2021-03-11 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Melanoma
Keywords: Precision radiation; PD-1 inhibitor; SBRT; Immune Checkpoint Inhibitor
MeSH Terms: conditions — Melanoma | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Phase II open-label multicenter trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Precision Radiation (SBRT) (Experimental): Precision radiation of melanoma metastases
  Interventions: Radiation: Precision Radiation (SBRT)

INTERVENTIONS:
Radiation: Precision Radiation (SBRT) — Precision radiation of melanoma metastases

SUMMARY:
To evaluate tumor response, survival and adverse effects after precision radiotherapy (SBRT) in melanoma patients with ongoing PD-1 inhibitor treatment that have tumor progression.

DETAILED DESCRIPTION:
A phase II open-label multicenter trial evaluating response rate (RR) in patients receiving precision radiation (SBRT) to melanoma metastasis that have progressed on PD-1 inhibitor therapy. Patients will continue on PD-1 inhibitor therapy (pembrolizumab or nivolumab) for up to one year after completed precision radiation and will be followed-up for 24 months or until disease progression or death. The primary endpoint of the study is overall response rate (ORR) in non-irradiated lesions. The study will be conducted according to Simon´s two Stage minimax Design. Patients will be enrolled in two batches, first consisting of 13 patients. If no objective responses (complete response (CR) or partial response (PR)) are reported after the first stage, the study is interrupted early for futility. When the 13th patient is recruited, if there is at least one objective response in patient´s non-irradiated lesion(s), the recruitment can proceed into second stage. 14 more patients will then be included up to a total of 27 patients to determine ORR along with the 95% confidence interval. The test result is considered positive when at least 15% of the patients have a confirmed objective response.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above
2. ECOG performance status of 0-1
3. Signed and dated written informed consent before the start of specific protocol procedures.
4. Patient has initiated PD-1 inhibitor treatment (alone or in combination with CTLA-4 inhibitor) as the first line of therapy for unresectable metastatic cutaneous melanoma and been on the treatment for at least 3 months and progressed on the treatment. Patients with primary or secondary resistance to the PD-1 inhibitor treatment will be included. Progression is defined as at least 30% enlargement of at least one metastasis or appearance of new metastasis. A fine-needle aspiration (FNA) biopsy from a progressing lesion or a new lesion is recommended to confirm the presence of viable tumor cells.
5. Patients on adjuvant treatment with PD-1 inhibitors that during the treatment develop unresectable biopsy confirmed metastases can also be included in the study.
6. Have at least one new or progressing lesion safely amenable to irradiation in the opinion of the treating radiation oncologist AND at least one, not-to-be-irradiated new or progressing lesion measurable by CT or MRI per RECIST 1.1 criteria where up to four radiation target fields are allowed
7. No contraindication for continuing immunotherapy after the radiotherapy intervention

Exclusion Criteria:

1. Inability to understand given information or undergo study procedures according to protocol
2. Pregnant or breast-feeding. Patients must agree to use safe contraception during and for 3 months after study treatment.
3. A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 30 days before start of study treatment. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted.
4. Has an active infection requiring systemic therapy.
5. Concomitant therapy with any anti-tumor medications, other than PD-1/CTLA-4 inhibitors or 30 days before and after treatment in this trial.
6. Prior radiotherapy preventing the study intervention with precision radiotherapy
7. Location, size or number of metastases is deemed as excessive or not appropriate for precision radiotherapy
8. Central nervous system (CNS) metastases at baseline, with the exception of those subjects who have previously-treated CNS metastases (surgery ± radiotherapy, radiosurgery, or gamma knife) and who meet both of the following criteria: a) are asymptomatic and b) have no requirement for steroids or anticonvulsants.
9. Prior malignancy. Subjects who have had another malignancy should be disease-free for 5 years, or should have a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) in non-irradiated lesions | From date of precision radiation start until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 24 months
  Overall response rate (ORR) in non-irradiated lesions according to RECIST 1.1

SECONDARY OUTCOMES:
Median PFS (months) | 6 and 12 months
  Median PFS (months) at 6 and 12 months according to RECIST 1.1
PFS rate (%) | 6 and 12 months
  PFS rate (%) at 6 and 12 months according to RECIST 1.1
Median OS (months) | 6 and 12 months
  Median OS (months) at 6 and 12 months according to RECIST 1.1
Response rate (RR) in the patient's irradiated lesions | From radiation start to end of follow-up, progression or death (3, 6, 9, 12, 15, 18, 21, 24 months)
  Response rate (RR) in the patient's irradiated lesions according to RECIST 1.1
Rate and type of AEs and SAEs on patient level | From precision radiation start to end of follow-up, progression or death, up to 24 months
  Adverse Events and Serious Adverse Events

OTHER OUTCOMES:
Exploratory outcome measure: Predictive biomarkers | From date of diagnosis until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 24 months
  Translational research to investigate predictive biomarkers based on sequential tumor biopsies and/or fine needle tumor aspirations and blood

CONTACTS AND LOCATIONS:
Overall Officials: Signe Friesland, MD, PhD, Study Director — Karolinska University Hospital
Locations (1):
- Division of Head-Neck, Lung and Skin cancers, Theme Cancer, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No